CLINICAL TRIAL: NCT05364931
Title: A Phase II Randomized, Double-blind, Placebo-controlled, Proof-of-Concept Study to Evaluate the Safety and Efficacy of Cotadutide in Participants With Non-cirrhotic Non-alcoholic Steatohepatitis With Fibrosis
Brief Title: A Study to Evaluate the Safety and Efficacy of Cotadutide Given by Subcutaneous Injection in Adult Participants With Non-cirrhotic Non-alcoholic Steatohepatitis With Fibrosis
Acronym: PROXYMO-ADV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5671C00006; 2021-005484-53 (EudraCT Number)
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Non-cirrhotic Non-alcoholic Steatohepatitis With Fibrosis
Keywords: NASH; fatty liver disease; non-alcoholic fatty liver; NAS; liver fibrosis; Non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cotadutide 300μg (Experimental)
  Interventions: Drug: Cotadutide
- Placebo 300μg (Placebo Comparator)
  Interventions: Drug: Placebo
- Cotadutide 600μg (Experimental)
  Interventions: Drug: Cotadutide
- Placebo 600μg (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cotadutide — Cotadutide administered subcutaneously once daily
  Arms: Cotadutide 300μg; Cotadutide 600μg
Drug: Placebo — Placebo administered subcutaneously once daily
  Arms: Placebo 300μg; Placebo 600μg

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of cotadutide in participants with non-cirrhotic NASH with fibrosis.

DETAILED DESCRIPTION:
A Phase 2, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of two different doses of cotadutide at 300 and 600 μg in participants with non-cirrhotic non-alcoholic steatohepatitis with fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Males and female participants ≥ 18 to ≤ 75 years of age (inclusive) at the time of signing the informed consent.
3. Histologically confirmed non-alcoholic steatohepatitis (NASH) per NASH Clinical Research Network (CRN) criteria as diagnosed by histology from a liver biopsy performed ≤ 180 days from randomization and fulfilling all of the following histological criteria:

   1. NAS (Non-alcoholic Fatty Liver Disease Activity Score) ≥ 4 with a score of ≥ 1 for each component: steatosis, lobular inflammation, and ballooning
   2. Presence of fibrosis stage F2 or F3
4. Women of childbearing potential, non-pregnant and nonbreastfeeding and using appropriate birth control to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study intervention.

Exclusion Criteria:

1. Chronic liver disease of other etiologies.
2. History of cirrhosis and/or hepatic decompensation, including evidence of portal hypertension (e.g. low platelet count, splenomegaly, ascites, history of hepatic encephalopathy, esophageal varices, or variceal bleeding).
3. Clinically significant cardiovascular or cerebrovascular disease within 90 days prior to screening, including but not limited to, myocardial infarction, acute coronary syndrome, unstable angina pectoris, transient ischemic attack, or stroke, or participants who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 90 days or who are due to undergo these procedures at the time of screening
4. History of malignant neoplasms within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or any in situ carcinoma.
5. Participation in another clinical study with an investigational product administered within the last 30 days or 5 half-lives of the therapy (whichever is longer) at the time of screening or the time of the historical biopsy or concurrent participation in another interventional study of any kind or prior randomization in this study.
6. Severe allergy/hypersensitivity to any of the proposed study treatments or excipients
7. Contraindication to liver biopsy (eg, bleeding diathesis, such as hemophilia, suspected hemangioma, or suspected echinococcal infection) or inability to safely obtain a liver biopsy as determined by the investigator
8. Severely uncontrolled hypertension defined as SBP ≥ 180 mmHg or DBP ≥ 110 mmHg on the average of 2 seated BP measurements after being at rest for at least 10 minutes at screening or randomization 9 Any positive results for human immunodeficiency virus infection, positive results for hepatitis B surface antigen or hepatitis C antibody test along with a positive HCV RNA test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (101):
- United States (26):
  - Research Site, Tucson, Arizona
  - Research Site, Canoga Park, California
  - Research Site, Gilroy, California
  - Research Site, Sacramento, California
  - Research Site, Englewood, Colorado
  - Research Site, Bradenton, Florida
  - Research Site, Homestead, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Munster, Indiana
  - Research Site, Houma, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Ann Arbor, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Lawrence, New Jersey
  - Research Site, Warren Township, New Jersey
  - Research Site, Morehead City, North Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Lewisville, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
- Research Site, CABA, Argentina
- Australia (5):
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Meadowbrook
  - Research Site, Melbourne
  - Research Site, Westmead
- Research Site, Vienna, Austria
- Canada (2):
  - Research Site, London, Ontario
  - Research Site, Terrebonne, Quebec
- France (2):
  - Research Site, Montpellier
  - Research Site, Paris
- Germany (2):
  - Research Site, Dresden
  - Research Site, Konstanz
- Greece (2):
  - Research Site, Athens
  - Research Site, Ioannina
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (6):
  - Research Site, Catania
  - Research Site, Foggia
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, San Giovanni Rotondo
- Japan (15):
  - Research Site, Chiba
  - Research Site, Fukui-shi
  - Research Site, Gifu
  - Research Site, Hiroshima
  - Research Site, Kawasaki-shi
  - Research Site, Kure-shi
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Takasaki-shi
  - Research Site, Toon-shi
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Malacca
  - Research Site, Seremban
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Grafton
- Research Site, Plumstead, South Africa
- South Korea (4):
  - Research Site, Busan
  - Research Site, Gangwon-do
  - Research Site, Junggu
  - Research Site, Seoul
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Almería
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Istanbul
- United Kingdom (8):
  - Research Site, Aberdeen
  - Research Site, Glasgow
  - Research Site, Ipswich
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Preston
  - Research Site, Rochdale
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5671C00006&attachmentIdentifier=ab9ab43f-7d52-4826-b285-72457171d41c&fileName=D5671C00006_Redacted_CSP.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5671C00006&attachmentIdentifier=1a7fca5f-0c40-449c-9b26-d1bec5b2b93e&fileName=D5671C00006_Redacted_SAP.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5671C00006&attachmentIdentifier=dde044fc-40da-4b3d-8a06-31550cf76396&fileName=D5671C00006_Redacted_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Cotadutide 300 ug: Cotadutide 300 ug QD
- Cotadutide 600 ug: Cotadutide 600 ug QD
- Placebo 600 ug: Placebo 600 ug QD
- Placebo 300 ug: Placebo 300 ug QD
Period: Overall Study
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo 600 ug | Placebo 300 ug
Started | 17 | 18 | 9 | 10
Completed | 14 | 14 | 5 | 8
Not Completed | 3 | 4 | 4 | 2
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 2
Not completed — study terminated by sponsor (reason as collected in database, study was not terminated) | 0 | 1 | 0 | 0
Not completed — Discontinued | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Although there are two placebo arms for blinding purposes, the safety and efficacy analyses in the (abbreviated) CSR pooled the two placebo arms and analyzed them as a single group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo 600 ug | Placebo 300 ug | Total
Number analyzed (Participants) | 17 | 18 | 9 | 10 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean(standard Deviation) | 54.4 (12.4) | 53 (12.6) | 56.4 (9.4) | 56.9 (11.6) | 54.7 (11.7)
Age, Customized [Number; unit: Participants] — Population: The full analysis set population
  Participants
    >= 65 years | 4 | 4 | 2 | 3 | 13
    >=50 - <65 years | 7 | 7 | 5 | 4 | 23
    < 50 years | 6 | 7 | 2 | 3 | 18
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The full analysis set population
  Participants
    Female | 11 | 10 | 6 | 4 | 31
    Male | 6 | 8 | 3 | 6 | 23
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The full analysis set population
  Participants
    American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
    Asian | 5 | 9 | 2 | 2 | 18
    Black or African American | 0 | 1 | 0 | 0 | 1
    Multiple | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Not Reported | 1 | 0 | 0 | 0 | 1
    Other | 0 | 0 | 0 | 0 | 0
    White | 11 | 8 | 6 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs).
Description: To assess safety and tolerability of Cotadutide. Occurrence of AEs and serious AEs, including AEs leading to dose reduction, and AEs of special interest.
Time Frame: First dose on Day 1 until the follow-up period, 28 days post last dose, up to approximately 52 weeks.
Population: Although there are two placebo arms for blinding purposes, the safety, immunogenicity, and efficacy analyses in the (abbreviated) CSR pooled the two placebo arms and analyzed them as a single group as prespecified in the SAP.
Measure: Count of Participants; unit: Participants
Groups:
- Cotadutide 600 ug: Cotadutide 300 ug QD
- Placebo: Placebo 300 ug or 600 ug QD
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo
Number analyzed (Participants) | 17 | 18 | 19
Participants | 16 | 16 | 13

2. Primary Outcome: Number of Participants With Abnormal Vital Signs.
Description: To assess safety and tolerability of Cotadutide.
Time Frame: First dose on Day 1 until the follow-up period, 28 days post last dose, up to approximately 52 weeks.
Population: Although there are two placebo arms for blinding purposes, the safety and efficacy analyses in the (abbreviated) CSR pooled the two placebo arms and analyzed them as a single group as prespecified in the SAP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo
Number analyzed (Participants) | 17 | 18 | 19
Participants | 13 | 14 | 17

3. Primary Outcome: Number of Participants With Abnormal Laboratory Assessments
Description: To assess safety and tolerability of Cotadutide.
Time Frame: First dose on Day 1 until the follow-up period, 28 days post last dose, up to approximately 52 weeks.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo
Number analyzed (Participants) | 17 | 18 | 19
Participants | 16 | 17 | 19

4. Primary Outcome: Number of Participants With Treatment Emergent Abnormality in 12-lead Electrocardiogram (ECG).
Description: To assess safety and tolerability of Cotadutide.
Time Frame: First dose on Day 1 until the follow-up period, 28 days post last dose, up to approximately 52 weeks.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo
Number analyzed (Participants) | 17 | 18 | 19
Participants | 4 | 2 | 6

5. Primary Outcome: Number of Treatment-induced Anti-Drug Antibody (ADA) Participants
Description: To assess the immunogenicity of Cotadutide
Time Frame: First dose on Day 1 until the follow-up period, 28 days post last dose, up to approximately 52 weeks.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo
Number analyzed (Participants) | 17 | 18 | 19
Participants | 7 | 11 | 0

6. Primary Outcome: Titer of Treatment-induced Anti-Drug Antibody (ADA)
Description: To assess the immunogenicity of cotadutide. Titers represent a dilution and are therefore unitless. Summary statistics are based on the maximum observed titer for each ADA positive subject within the time frame.
Time Frame: From first dose on Day 1 until the follow-up period, 28 days post last dose (from randomization up to approximately 52 weeks).
Measure: Median (Full Range); unit: titer
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug
Number analyzed (Participants) | 17 | 18
titer | 240 [15 to 7680] | 60 [15 to 240]

ADVERSE EVENTS:
Time Frame: From first dose on Day 1 up to approximately 52 weeks.
Groups:
- Cotadutide 300 ug; Cotadutide 600 ug; Placebo 600 ug; Placebo 300 ug: Description (Arm-group)
Arm/Group | Cotadutide 300 ug | Cotadutide 600 ug | Placebo 600 ug | Placebo 300 ug
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/18 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/18 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 16/17 | 17/18 | 5/9 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cotadutide 300 ug (N=17) | Cotadutide 600 ug (N=18) | Placebo 600 ug (N=9) | Placebo 300 ug (N=10)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pacemaker generated arrhythmia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cotadutide 300 ug (N=17) | Cotadutide 600 ug (N=18) | Placebo 600 ug (N=9) | Placebo 300 ug (N=10)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (7) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 9 (14) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 6 (8) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT05364931/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT05364931/SAP_001.pdf